CLINICAL TRIAL: NCT02271763
Title: A Descriptive Study Comparing a Horizontal Ultrasound Technique With a Palpation Technique for Localising the Cricothyroid Membrane in an Obstetric Population.
Brief Title: Comparing a Horizontal Ultrasound Technique With a Palpation Technique for Localising the Cricothyroid Membrane
Acronym: CTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double
Other Study IDs: H14-01177; CW14-0188 (Other: Children's & Women's Health Centre of BC)
Record Dates: First submitted 2014-09-26; First posted 2014-10-22 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Airway Identification
Keywords: cricothyroid membrane; ultrasound
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palpating neck (Active Comparator): Subjects will have their neck palpated by an anesthesiologist to locate their cricothyroid membrane
  Interventions: Other: ultrasound
- Ultrasound neck (Experimental): Subjects will have their neck scanned with ultrasound by an anesthesiologist to locate their cricothyroid membrane
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — subjects' neck will be scanned using ultrasound

SUMMARY:
The investigators will be comparing a traditional palpation (feeling) technique with an ultrasound technique for finding a specific part of the neck.

DETAILED DESCRIPTION:
This study compares a traditional palpation (feeling) technique with an ultrasound technique for finding a specific part of the neck. Finding this part of the neck is important for anesthesiologists in emergencies and can sometimes be difficult. We would like to determine if using ultrasound is easier and more reliable than examining the neck by hand. Newer methods using ultrasound have not been studied in detail in the pregnant population.

This study aims to describe a simple technique for identifying the cricothyroid membrane. The secondary aim is to determine how ultrasound compares to palpation in pregnant women at term.

ELIGIBILITY:
Inclusion Criteria:

* term pregnancy
* 19yrs and older

Exclusion Criteria:

* preterm pregnancy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Airway localization | 10 minutes
  Subjects necks' will be palpated and then scanned using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Simon Massey, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada